CLINICAL TRIAL: NCT02207712
Title: Noctura400 Treatment for Diabetic Retinopathy: Pilot Study to Demonstrate and Evaluate the Care Pathway for National Health Service (NHS) Adoption
Brief Title: Noctura400 Treatment for Diabetic Retinopathy (CANDLE)
Acronym: CANDLE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Major protocol deviations compromised the study.
Sponsor: PolyPhotonix Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PPX-2014-004
Record Dates: First submitted 2014-07-24; First posted 2014-08-04 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Diabetic Macular Oedema
Keywords: Diabetes; Macular Oedema; Diabetic retinopathy; Noctura
MeSH Terms: conditions — Diabetes Mellitus; Macular Edema; Diabetic Retinopathy | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Arm (Active Comparator): Those receiving only their prescribed ranibizumab treatment only
  Interventions: Drug: Ranibizumab
- Intervention Arm (Experimental): Noctura 400 Eye Mask in conjunction with their prescribed ranibizumab treatment.
  Interventions: Device: Noctura 400 Eye Mask; Drug: Ranibizumab

INTERVENTIONS:
Device: Noctura 400 Eye Mask — The intervention is the wearing of the eye mask
  Other Names: Noctura400
  Arms: Intervention Arm
Drug: Ranibizumab — Standard ranibizumab treatment only
  Other Names: Those receiving their standard ranibizumab treatment only

SUMMARY:
In this study, the investigators aim to use light masks (Noctura 400) to test the hypothesis that preventing the dark adaptation and associated hypoxia of the rods in the eye could in turn prevent or halt the progression of centre-involving Diabetic Macular Oedema (DMO). DMO is a devastating disease that is the most common cause of registerable blindness in the working age-group in the United Kingdom (UK)

This is a multi-centred randomised controlled trial involving 240 patients. Post randomization, participants in the intervention arm will wear the Noctura 400 Light Mask at night for 48 weeks in conjunction with their routine, prescribed treatment of intravitreal (eye) ranibizumab. Those in the standard arm will receive their routine, prescribed ranibizumab treatment only.

The primary objective is to determine whether utilizing the Noctura 400 Light Mask at night reduces the number of intravitreal injections of ranibizumab required by patients undergoing such a course for the treatment of DMO.

DETAILED DESCRIPTION:
Diabetes is regarded by the World Health Organisation (WHO) as a global epidemic, with the global diabetic population anticipated to exceed 500 million by 2020. In the UK there are over 3.5 million people who have diabetes with a growth rate exceeding 150,000 people per year. Diabetic Retinopathy (DR) is the most common complication of diabetes, and the most common cause of sight threatening retinopathy is Diabetic Macular Oedema (DMO).

This condition is characterised by leakage of fluid from compromised blood vessels in the central retina and 240,000 (8%) people with diabetes in the UK have clinically significant DMO, and 100,000 people with DMO have visual impairment. DMO is the most common cause of registerable blindness in the working age-group in the UK. The Diabetic Eye Screening Programme (DESP) annually photographs 3 million people with diabetes at a cost of £65 million to ensure early diagnosis of these sight threatening complications. All patients with diabetic maculopathy are referred to the Hospital Eye Service (HES).

Clinically significant macular oedema requires treatment. Non-central oedema is usually kept under close monitoring or laser treatment is advocated. Centre involving macular oedema is usually treated with intravitreal injections of inhibitors of Vascular Endothelial Growth Factor (anti-VEGF). Whilst laser treatment can reduce the risk of moderate visual loss by 50%, it is not effective in restoring best corrected visual acuity (BCVA) and has significant, quality of life impacting side effects. The anti-VEGF treatments are costly and cause significant burden to patients, their care-givers and the healthcare system.

A patient with DR never leaves the HES. With diabetes on the rise the cost of care for this ever increasing population is growing year on year. This is putting immense strain on the resources and budgets of the healthcare system.

In this trial the investigators will explore the health and economic impact of a new, novel therapy for DMO provided by the Noctura 400 Light Mask. The Light Mask provides a non-invasive, light therapy that can be administered at home by the patients themselves. If successful, the introduction of Noctura 400 Light Mask treatment could bring significant benefits to both patients and the healthcare system.

This trial has been designed as a randomised control trial to allow the direct assessment of the Noctura 400 treatment based on a comparison with a control arm of patients not receiving this treatment. All participants in the trial will be due to undergo their first year of a course of intravitreal injection of an anti-VEGF drug known as ranibizumab. Those in the treatment arm will, in addition to this course of injections, wear the Noctura 400 Light Mask each night for 48 weeks. Those in the standard, or control, arm will receive their course of injections only.

The study will involve 240 participants who have been diagnosed with clinically significant DMO and referred to the Hospital Eye Service (HES) for injections. The current threshold for referral is central retinal thickening of 400um or greater. Once in the HES, potential participants will be assessed for eligibility in clinic. These eligibility tests will form the future participant's "baseline visit". If eligible, patients will be invited to participate in the study. The eligibility assessment requires no further tests to those required by the routine care pathway.

After gaining informed consent, eligible and consenting participants will then be randomised into either the intervention arm (those wearing the Noctura 400 Light Mask each night in conjunction with their routine injections) or a standard arm (those receiving their injections only) and will then be invited back to clinic to begin their allocated therapy.

At the first trial visit, those in the intervention arm will be given the Noctura 400 Light Mask to take away with them and instructed how to use it. The Noctura 400 is powered and programmed to last for precisely 12 weeks. Participants will be provided with a replacement mask at appropriate appointments to ensure continuous treatment.

At each and every appointment all participants will undergo Optical Coherence Tomography (OCT) measurements (for assessment of disease progression) and visual acuity (VA) tests. For the first three visits all participants will be given intravitreal injections, following this, participants in both arms will be given injections at appointments only if required based on the results of the OCT and VA tests. Medical history, concomitant medications and adverse events will be recorded at each visit. At weeks 0,12 and 48 patients will fill out insomnia and sleepiness and quality of life questionnaires.

The Noctura 400 has the ability to sense and record when it has been used as a direct measure of compliance. Sleep Mask data will be collected at weeks 12,24,26 and 48. If compliance is low this will be discussed with the participant with the aim of increasing compliance. If at any point during the trial the Noctura 400 Light Mask appears faulty it will be returned for analysis and replaced.

The trial ends at the patient's last visit after 48 weeks of use. Participants will return their Noctura 400 Light Masks for analysis and then patients in both arms are free to continue their routine injections as prescribed by the current care pathway. Participants will be made aware at the time of consenting that the Noctura 400 Light Mask will not be available within the NHS at the end of the trial, but that the manufacturer intends for the device to be available to purchase privately

ELIGIBILITY:
Inclusion Criteria:

i. Subjects of either sex aged 18 years or over. ii. Diagnosis of diabetes mellitus (type 1 or type 2). iii. Presence of clinically significant centre-involving macular oedema resultant from DR of ≥400µm (CST/CMT as measured by OCT, and is listed for ranibizumab therapy in the study eye.

Exclusion Criteria:

Any potential participant will be excluded if they have:

i. Received any previous anti-VEGF/steroid intravitreal injections in the study eye in the last 6 months.

ii. Presence of proliferative diabetic retinopathy (PDR) at screening.

iii. Significant systemic diseases know to affect visual function, other than diabetes (e.g. Parkinson's disease or Alzheimer's disease).

iv. History of relevant sleeping disorders/insomnia .

v. A condition that would preclude participation in the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2023-08 (Actual); Study Completion 2023-08 (Actual)

PRIMARY OUTCOMES:
The number of intravitreal injections of ranibizumab required by each study eye at 48 weeks | 48 Weeks

SECONDARY OUTCOMES:
Mean difference from baseline Central sub-field thickness at 48 Weeks | 48 Weeks
Mean difference from baseline visual acuity at 48 weeks. | 48 Weeks
Mean difference in utility (quality of life). | Baseline, 12 and 48 weeks
Difference in the number of ranibizumab injections received by patients who have received at least three injections. | Between weeks 12 and 48
Change in Central sub-field thickness over time | 12, 24,36 and 48 Weeks
Pattern of injections given over the period of 48 weeks in both arms. | 48 weeks
Adverse events rates | 48 months

OTHER OUTCOMES:
Compliance of wearing the mask | 48 weeks
Changes in sleep pattern. | 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Martin Holland, Study Chair — PolyPhotonix Medical; Ulrich Meyer-Bothling, Principal Investigator — Ashford & St Peters Hospitals NHS Trust
Locations (18):
- United Kingdom (18):
  - Royal Berkshire NHS Foundation Trust, Reading, Berkshire
  - Hitchingbrooke Healthcare NHS Trust, Huntingdon, Cambridgeshire
  - Peterborough and Stamford Hospitals NHS Foundation Trust, Peterborough, Cambridgeshire
  - South Tees Hospitals NHS Foundation Trust, Middlesbrough, Cleveland
  - Royal Cornwall Hospitals NHS Trust, Truro, Cornwall
  - Colchester Hospital University NHS Foundation Trust, Colchester, Essex
  - Glouchestershire Hospitals NHS Foundation Trust, Cheltenham, Glouchestershire
  - Basingstoke and North Hampshire NHS Foundation Trust, Basingstoke, Hampshire
  - North Lincolnshire and Goole NHS Trust, Scunthorpe, Lincolnshire
  - James Paget University Hospital NHS Foundation Trust, Great Yarmouth, Norfolk
  - Norfolk and Norwich University Hospitals NHS Foundation Trust, Colney, Norwich Norfolk
  - Oxford Radcliffe Hospitals NHS Trust, Headington, Oxford Oxfordshire
  - Yeovil District Hospital NHS Foundation Trust, Yeovil, Somerset
  - Ashford & St Peters Hospitals NHS Foundation Trust, Chertsey, Surrey
  - Royal Surrey County Hospital, Guildford, Surrey
  - Mid Yorkshire Hospitals NHS Trust, Wakefield, West Yorkshire
  - Great Western Hospital, Swindon, Wiltshire
  - Plymouth Hospitals NHS Trust, Plymouth

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor Website — http://www.polyphotonix.com